CLINICAL TRIAL: NCT06367140
Title: Effects of Electromyography-Triggered Constraint-Induced Movement Cycling Therapy on Patients With Chronic Stroke: A Randomized Controlled Trial
Brief Title: Effects of Electromyography-Triggered Constraint-Induced Movement Cycling Therapy on Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Collaborators: Seoul National University Hospital (Other); Kyungdong University (Other)
Responsible Party: Principal Investigator, Changho Song, professor, Sahmyook University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2021-06-001-002
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Postural balance; Electromyography; Muscle Strength; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluators were blinded to the intervention details of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- constraint-induced movement therapy groups (Experimental): The device utilized EMG sensors to collect signals from the leg muscles, which then controlled the cycling motion. This group underwent specific training sessions designed to enhance muscle activation on the affected side by inducing voluntary contractions through cycling, with the aim of improving muscle strength, balance, and activities of daily living. The sessions included a structured regimen of warm-up, active cycling with therapist-guided acceleration based on muscle activation, and cool-down periods, conducted under supervision for safety and effectiveness.
  Interventions: Device: EMG-triggered CIMCT device
- general cycling training groups (Sham Comparator): This group followed a similar session structure to the CIMCT group, including warm-up, cycling at a comfortable pace, and cool-down phases, but without the targeted muscle activation component.
  Interventions: Device: general cycling training

INTERVENTIONS:
Device: EMG-triggered CIMCT device — The study tested an EMG-triggered CIMCT device for stroke rehab, involving EMG sensors, a stationary bike, and a control unit displaying muscle activity. The protocol included warm-up, therapist-guided exercises, and cool-down, performed under supervision.
  Arms: constraint-induced movement therapy groups
Device: general cycling training — The training aimed to improve overall physical fitness and potentially aid in stroke recovery through regular cycling activity, conducted under supervision to ensure participant safety and adherence to the protocol.
  Arms: general cycling training groups

SUMMARY:
The study investigates the potential of Electromyography (EMG)-triggered Constraint-Induced Movement Cycling Therapy (CIMCT) versus General Cycling Training (GCT) to enhance balance, strength, and daily activities in chronic stroke patients. Over a period of four weeks, this single-blind randomized controlled trial aims to explore how these interventions can assist in stroke rehabilitation. The research has been approved by the Ethics Committee of Kyungdong University and adheres to the ethical standards laid out in the Declaration of Helsinki.

DETAILED DESCRIPTION:
This research evaluates the effectiveness of EMG-triggered CIMCT in improving balance, lower extremity strength, and activities of daily living (ADLs) for chronic stroke patients with hemiplegia, a condition typically resulting from a stroke. The study's scope includes:

Duration and Type: A four-week, single-blind randomized controlled trial. Participants: Chronic stroke patients diagnosed with stroke-induced hemiplegia for more than six months, possessing specific levels of cognitive and motor recovery.

Interventions: Participants are randomly assigned to one of two groups:

CIMCT Group: Utilizes an EMG-triggered Constraint-Induced Movement Therapy device designed to engage the affected lower extremity actively.

GCT Group: Engages in activity using a standard stationary bicycle without EMG facilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stroke-induced hemiplegia
* Diagnosed with stroke for more than 6 months
* Achieving a minimum score of 24 points on the Mini-Mental State Examination
* Demonstrating motor recovery at or above level 3 according to the Brunnstrom stages

Exclusion Criteria:

* Individuals with neurological damage unrelated to their stroke
* Orthopedic issues such as fractures or peripheral nervous system damage in the lower limbs
* Visual or auditory impairments
* Those who had experienced more than one stroke
* Those with less than an 80% participation rate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | baseline-4weeks
  A manual muscle tester (Model 01163, Lafayette, USA, 2003) was used to evaluate lower extremity muscle strength in this study. The knee extensors, knee flexors, dorsiflexors, and plantar flexors, which are primarily responsible for the pedaling motion, were assessed. Moreover, both sides were evaluated.
Static Balance | baseline-4weeks
  This study utilized a commercially available GB300 (Metitur Ltd., Jyvaskyla, Finland) posture measurement system for posture measurement, which included a movable triangular-shaped platform and a ruler that displayed the position of the feet. The aforementioned system was useful for analyzing balance problems and the effectiveness of rehabilitation. The posture management system is also commonly used to assess balance ability in athletes, older individuals, patients with stroke, and patients with hemiplegia. The sampling frequency was set at 50 Hz. The participants stood with their eyes open and facing forward for 30 s while fixed to the equipment; this was repeated three times. Subsequently, they stood in the same position with their eyes closed and facing forward for 30 s for three additional measurements.
Timed Up and Go (TUG) | baseline-4weeks
  The Timed up-and-go (TUG) test was used to assess the balance ability in this study. In the test, the participant sits in a chair with armrests, rises from the chair at the same time as the word "start" is spoken, walks at the most stable and comfortable speed to a point 3 m in front of them, and then returns and measures the time to sit down in the chair. It has a high intra-rater reliability (r=.99) and inter-rater reliability (r=.98). The raters performed three measurements using a stopwatch and recorded the average value.
Berg Balance Scale | baseline-4weeks
  The Berg Balance Scale is used to assess functional balance in a wide range of participants, including older individuals at a high risk of falling and patients with acute and chronic diseases. Moreover, Berg Balance Scale is a functional balance test method that considers three aspects of functional balance: postural maintenance, postural control by manual exercise, and response to external perturbations. these activities are scored from 0 to 4, with 0 being the worst and 4 being the best performance of independent tasks. The maximum total score is 56 points. A lower score suggests impaired stability.
Functional Reach Test (FRT) | baseline-4weeks
  The functional reach test (FRT) assesses the limits of physical stability and measures dynamic balance and flexibility while the participant performs a functional task. The FRT measures the maximum distance a participant can extend their arm forward from a standing position while maintaining fixed support. The distance was measured in centimeters using a Laser Rangefinder (DLE50, BOSCH, Germany). The results represented the averages of three consecutive measurements. The reliability of this test was 0.89.
Modified Barthel Index (MBI) | baseline-4weeks
  The modified Barthel index (MBI) developed by was used to measure the performance of daily living behaviors. The MBI consists of 10 items: self-care, bathing, feeding, climbing stairs, dressing, bowel control, bladder control, walking, and transferring. The scoring system ranged from 5 to 15, with a score of 100 if all items could be performed completely independently. The inter-rater reliability was 0.93-0.98, and the Cronbach's alpha value was 0.84.

CONTACTS AND LOCATIONS:
Overall Officials: Jaemyoung Park, Ph.D., Study Chair — Sahmyook University; Jung hyun Kim, prof, Study Director — Seoul National University Hospital; Kyeongjin Lee, prof, Study Director — Kyungdong University; Changho Song, prof, Principal Investigator — Sahmyook University
Locations (1):
- Department of Physicla Therapy, Sahmyook University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No